CLINICAL TRIAL: NCT05428488
Title: Efficacy of a Sequential Treatment Strategy in Rheumatoid Arthritis. A Randomized Controlled Trial With an Independent Efficacy Assessor.
Brief Title: Efficacy of a Sequential Treatment Strategy in Rheumatoid Arthritis
Acronym: SEQUENS-RA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL21_0568
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; sequential therapeutic strategy; immunological remission; anti-TNF; abatacept
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Tumor Necrosis Factor Inhibitors

STUDY DESIGN:
Intervention Model Description: This study will include a 12 weeks non-randomized phase. This phase will include RA patients ACPA+ with insufficient response to cs DMARDs and eligible for TNF inhibitors. All included patients will receive TNF inhibitors subcutaneous for 12 weeks.
  At 12 weeks visit (W12), patients who have at least a moderate EULAR response (delta DAS28-CRP between and W0 and W12>0.6 and DAS28-CRP≤5.1 at W12) will be randomized with a 1:1 ratio in the sequential strategy arm or the control arm. Then, the randomized phase will be 36 weeks long.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): All included patients will receive TNF inhibitors subcutaneous for 12 weeks. In the experimental arm, a therapeutic sequential strategy will be proposed from W12 visit.
  At 12 weeks (W12), patients who have at least a moderate EULAR response (delta DAS28-CRP between W0 and W12>0.6 and DAS28-CRP≤5.1 at W12) will be randomized with a 1:1 ratio in the sequential strategy arm or the control arm.
  In the sequential strategy (experimental) arm, the 88 randomized RA patients will be switched to abatacept subcutaneous for 36 weeks.
  Interventions: Drug: Abatacept (W12-W48); Drug: TNF Inhibitor (W0-W12)
- Control (Active Comparator): All included patients will receive TNF inhibitors subcutaneous for 12 weeks. In the control group, the 88 randomized RA patients will be treated with TNF inhibitor subcutaneous for another 36 weeks (from W12 visit).
  In case of insufficient response to a first TNF inhibitor at 24 or 36 weeks, a second TNF inhibitor will be proposed.
  Interventions: Drug: TNF Inhibitor (W12-W48); Drug: TNF Inhibitor (W0-W12)

INTERVENTIONS:
Drug: Abatacept (W12-W48) — The experimental strategy will evaluate abatacept 125 mg/week following 12 weeks of anti-TNF prescribed in usual care. Concomitant treatment with stable doses of csDMARD, non-steroidal anti-inflammatory drugs, analgesic agents, glucocorticoids (≤10 mg of prednisone or the equivalent per day), or a combination of these drugs will be permitted.
  Patients will continue to take methotrexate or leflunomide for the duration of the study.
  Arms: Experimental
Drug: TNF Inhibitor (W12-W48) — In the control group, the 88 randomized RA patients will be treated with TNF inhibitor subcutaneous for 36 weeks. In case of insufficient response to a first TNF inhibitor at 24 or 36 weeks, a second TNF inhibitor will be proposed.
  Arms: Control
Drug: TNF Inhibitor (W0-W12) — All included patients will receive TNF inhibitors subcutaneous for 12 weeks.

SUMMARY:
In rheumatoid arthritis (RA), the consensual 1st line conventional synthetic disease modifying antirheumatic drugs (csDMARD) of RA is methotrexate (MTX). In case of contra-indication or intolerance to MTX, leflunomide is an alternative. If the treatment target is not achieved with csDMARD strategy, addition of a biological DMARD (TNF inhibitors, anti-Interleukin 6 (anti-IL6)), abatacept, or rituximab) or a targeted synthetic (ts) DMARD (JAK inhibitors) is considered.

Current practice is to start a bDMARD (biologic Disease Modifying Antirheumatic Drugs) and especially TNF inhibitors (etanercept or monoclonal anti-TNF antibodies) with the benefit of hindsight. However, abatacept and TNF inhibitors have demonstrated similar efficacy in patients with insufficient response to csDMARD (AMPLE trial).

Although abatacept has shown a very good tolerance profile that might be superior to other bDMARDs rheumatologists might be reluctant to use it as a first line bDMARD as there is a belief of a slower efficacy compared to other bDMARDs or JAK inhibitors. Indeed, in real world study, compared to TNF inhibitors it seems that discontinuation of abatacept is more related to lack of effectiveness than safety issues.

Investigators have hypothesized that first rapidly controlling the inflammation phase, using TNF inhibitors followed by abatacept to induce an immunological remission would optimize response and tolerance of ACPA positive patients with RA. To demonstrate our hypothesis, the investigaors propose a randomized controlled trial with one arm receiving an induction therapy for 12 weeks with a TNF inhibitor followed by a cell-targeted bDMARD (abatacept) and the other arm, receiving TNF inhibitors.

DETAILED DESCRIPTION:
In rheumatoid arthritis (RA), the consensual 1st line conventional synthetic disease modifying antirheumatic drugs (csDMARD) of RA is methotrexate (MTX) (1). In case of contra-indication or intolerance to MTX, leflunomide is an alternative. If the treatment target is not achieved with csDMARD strategy, addition of a biological (b) DMARD (TNF inhibitors, anti-IL6, abatacept, or rituximab) or a targeted synthetic (ts) DMARD (JAK inhibitors) is considered.

Current practice is to start a bDMARD and especially TNF inhibitors (etanercept or monoclonal anti-TNF antibodies) with the benefit of hindsight. However, abatacept and TNF inhibitors have demonstrated similar efficacy in patients with insufficient response to csDMARD (AMPLE trial).

Although abatacept has shown a very good tolerance profile that might be superior to other bDMARDs rheumatologists might be reluctant to use it as a first line bDMARD as there is a belief of a slower efficacy compared to other bDMARDs or JAK inhibitors. Indeed, in real world study, compared to TNF inhibitors it seems that discontinuation of abatacept is more related to lack of effectiveness than safety issues.

This is the first study to propose a therapeutic sequential strategy with an induction therapy using a TNF inhibitor for 12 weeks to control inflammation followed by a cell-targeted biological DMARD targeting T cells (abatacept) in order to decrease auto-antibodies (rheumatoid factor and/or ACPA).

Presence of auto-antibodies (ACPA/RF) are predictive of better response to cell- targeted DMARDs.

In early AMPLE trial, RA patients ACPA+ with insufficient response to MTX were treated with abatacept or adalimumab. DAS28-CRP remission rates were 55% in abatacept group and 30% in adalimumab group.

Patients carrying the shared epitope (HLA-DR (Human Leucocyte Antigen-DR) alleles associated with RA), were also more likely to reach remission (DAS28-CRP<2.6) with abatacept (50%) than adalimumab (23%) at 24 weeks.

The clinical trial offered by investigateors here could change the paradigm in the strategy used in RA supporting the importance to first control inflammation environment in order to allow the cell-targeted bDMARDs to control immunological process which has been recently associated with a higher percentage of clinical remission.

To compare the percentage of remission (DAS28-CRP<2.6) obtained during the 36 weeks following randomization, with a sequential therapeutic strategy using abatacept versus a routine strategy continuing TNF inhibitors (TNFi), in ACPA positive RA patients responding to a first TNFi, initiated 12 weeks before randomization.

The primary endpoint will be analyzed with a generalized estimating equations (GEE) model for repeated data.

It is a multicentric, open label, randomized controlled trial comparing two different strategies of treatment with an independent efficacy assessor. For this clinical trial, to limit response bias, bDMARDs with a similar mode of administration (subcutaneous) are proposed.

In the experimental arm, a therapeutic sequential strategy will be proposed and in the control arm TNF inhibitors will be proposed for 48 weeks. All included patients will receive TNF inhibitors subcutaneous for 12 weeks. At 12 weeks (W12), patients who have at least a moderate EULAR response (delta DAS28-CRP between W0 and W12>0.6 and DAS28-CRP≤5.1 at W12) will be randomized with a 1:1 ratio in the sequential strategy arm or the control arm. In the sequential strategy arm, the 88 randomized RA patients will be switched to abatacept subcutaneous for 36 weeks. Patients who will withdraw abatacept during the follow-up will be considered as a failure.

In the control group, the 88 randomized RA patients will be treated with TNF inhibitor subcutaneous for another 36 weeks. In case of insufficient response to a first TNF inhibitor at 24 or 36 weeks, a second TNF inhibitor will be proposed. Anti-TNF drugs withdrawal will be considered as a failure. Steroids 0.1mg/kg/ day will be allowed but at stable dose 2 weeks before and with guided step-down strategy targeting withdrawal before 24 weeks following randomization. Clinical evaluation of disease activity using different scores (DAS28-ESR, CDAI, SDAI, Boolean criteria) and tolerance will be performed at all visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 or above
* Rheumatoid arthritis according to ACR-EULAR 2010 (American College of Rheumatology-European League Against Rheumatism)
* ACPA positive
* Under methotrexate or leflunomide treatment for at least 3 months
* DAS28-CRP>3.2 under methotrexate or leflunomide calculated with CRP dated less than 7 days from baseline
* Escape under synthetic background treatment defined by an elevation of C-reactive protein (CRP) (CRP> 5mg/L ) or Erythrocyte sedimentation rate (ESR) (for men: > age in years/2 ; for women: > age (+10) /2)) within the last 6 months before baseline
* Targeted DMARDs (biological and targeted synthetic DMARDs) naïve
* Indication for a TNF inhibitor

Exclusion Criteria:

* Subject unable to read or/and write
* Planned longer stay outside the region that prevents compliance with the visit plan
* Subject unable to sign informed consent form
* Subject not covered by public health insurance
* Dementia
* Fibromyalgia
* Contra-indications to TNF inhibitor and/or Abatacept
* Absence of tuberculosis screening in the previous 3 months before baseline
* Patient with untreated active tuberculosis
* Patient who cannot be followed during 48 weeks
* Drug addiction, addiction to alcohol
* Protected populations according to the French Public Health Code Articles L1121-5,6,8 (For example, pregnant, parturient or lactating women, prisoners, adults under guardianship or otherwise unable to consent).
* Women of child bearing potential, unless they are using an effective method of birth control
* Patient under law protection
* Prisoners
* Subject who are in a dependency or employment with the sponsor or the investigator
* Participation in another interventional clinical trial or administration of an investigational product within the last 4 weeks before the screening date
* Subject with moderate to severe heart failure (class 3 or class 4 cardiac disease as defined by the New York Heart Association Functional Classification)
* Patients had a history of chronic obstructive pulmonary disease (COPD) and heavy smoking
* Patients had a planned surgical procedure at least 30 days before the screening day
* Known allergy or intolerance to an anti-TNF therapy
* Hypersensitivity to the Abatacept or to any of its excipients
* Patient with untreated active hepatitis B
* Patient vaccinated with a live vaccine within 30 days prior to screening
* Patients with an Inflammatory Bowel Disease (IBD) (loss of chance if switching from an anti-TNF to abatacept)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in remission | 36 weeks following randomization
  Percentage of patients in remission defined by DAS28-CRP<2.6 score during the 36 weeks following randomization.
  Disease Activity Score-28 with C-Reactive Protein (DAS28-CRP) describes severity of rheumatoid arthritis using clinical and laboratory data, specifically CRP.
  It includes 4 variables (number of painful joints out of 28 joints, number of swollen joints out of 28 joints, global assessment of the disease by the patient on a Visual Analogue Scale (VAS), markers of inflammation : CRP)
  A DAS28-CRP score > 5.1 means high disease activity, DAS28-CRP < or = 3.2 indicates low disease activity, a DAS28-CRP < 2.6 indicates disease remission.

SECONDARY OUTCOMES:
percentage of patients in remission at 12 weeks after randomization (DAS28-ESR) | At 24 weeks visit (corresponding to 12 weeks after randomization)
  Percentage of patients in remission using definition : DAS28-ESR<2.6, at 12 weeks after randomization
  Disease Activity Score-28 with Erythrocyte Sedimentation Rate (DAS28-ESR) describes severity of rheumatoid arthritis using clinical and laboratory data, specifically ESR.
percentage of patients in remission at 12 weeks after randomization (CDAI) | At 24 weeks visit (corresponding to 12 weeks after randomization)
  Percentage of patients in remission using definition : CDAI≤2.8, at 12 weeks after randomization
  Clinical Disease Activity Index (CDAI) is a useful clinical composite score. It's the sum of 4 parameters : Swollen 28-Joint + Tender 28-Joint Count + Patient Global disease Activity + Evaluator's Global disease Activity.
  Remission is defined as an CDAI of ≤2.8, low disease activity as >2.8 and ≤10, moderate disease activity as >10 and ≤22 and high disease activity as >22.
percentage of patients in remission at 12 weeks after randomization (SDAI) | At 24 weeks visit (corresponding to 12 weeks after randomization)
  Percentage of patients in remission using definition : SDAI≤3.3, at 12 weeks after randomization
  Score Disease Activity Index (SDAI) is the sum of 5 parameters: the number of painful joints and synovitis (28 joints are tested) the global assessment of the patient and the therapist on a visual
percentage of patients in remission at 12 weeks after randomization (Boolean) | At 24 weeks visit (corresponding to 12 weeks after randomization)
  Percentage of patients in remission using definition: Boolean criteria, at 12 weeks after randomization Boolean criteria of remission are : number of tender and swollen joint, visual analogue scale for global health and CRP all ≤1
Percentage of patients in remission at 24 weeks after randomization (DAS28-ESR) | At 36 weeks visit (corresponding to 24 weeks after randomization)
  Percentage of patients in remission using definition : DAS28-ESR<2.6, at 24 weeks after randomization
Percentage of patients in remission at24 weeks after randomization (CDAI) | At 36 weeks visit (corresponding to 24 weeks after randomization)
  Percentage of patients in remission using definition : CDAI≤2.8, at 24 weeks after randomization
Percentage of patients in remission at 24 weeks after randomization (SDAI) | At 36 weeks visit (corresponding to 24 weeks after randomization)
  Percentage of patients in remission using definition : SDAI≤3.3, at 24 weeks after randomization
Percentage of patients in remission at 24 weeks after randomization (Boolean) | At 36 weeks visit (corresponding to 24 weeks after randomization)
  Percentage of patients in remission using definitions : Boolean criteria, at 24 weeks after randomization
Percentage of patients in remission at 36 weeks after randomization (DAS28-ESR) | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Percentage of patients in remission using definition : DAS28-ESR<2.6, at 36 weeks after randomization
Percentage of patients in remission at 36 weeks after randomization (CDAI) | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Percentage of patients in remission using definition : CDAI≤2.8, at 36 weeks after randomization
Percentage of patients in remission at 36 weeks after randomization (SDAI) | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Percentage of patients in remission using definition : SDAI≤3.3, at 36 weeks after randomization
Percentage of patients in remission at 36 weeks after randomization (Boolean) | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Percentage of patients in remission using definition : Boolean criteria at 36 weeks after randomization
Percentage of patients with low disease activity at 12 weeks after randomization (DAS28-ESR) | At 24 weeks visit (corresponding to 12 weeks after randomization)
  Percentage of patients in low disease activity using definition : 2.6≤DAS28-ESR≤3.2, at 12 weeks after randomization:
Percentage of patients with low disease activity at 12 weeks after randomization (DAS28-CRP) | At 24 weeks visit (corresponding to 12 weeks after randomization)
  Percentage of patients in low disease activity using definition : 2.6≤DAS28-CRP≤3.2, at 12 weeks after randomization
Percentage of patients with low disease activity at 12 weeks after randomization (CDAI) | At 24 weeks visit (corresponding to 12 weeks after randomization)
  Percentage of patients in low disease activity using definition : 2.8<CDAI≤10, at 12 weeks after randomization
Percentage of patients with low disease activity at 12 weeks after randomization (SDAI) | At 24 weeks visit (corresponding to 12 weeks after randomization)
  Percentage of patients in low disease activity using definition : 3.3<SDAI≤11, at 12 weeks after randomization
Percentage of patients with low disease activity at 24 weeks after randomization (DAS28-ESR) | At 36 weeks visit (corresponding to 24 weeks after randomization)
  Percentage of patients in low disease activity using definition: 2.6≤DAS28-ESR≤3.2, at 24 weeks after randomization
Percentage of patients with low disease activity at 24 weeks after randomization (DAS28-CRP) | At 36 weeks visit (corresponding to 24 weeks after randomization)
  Percentage of patients in low disease activity using definition : 2.6≤DAS28-CRP≤3.2, at 24 weeks after randomization
Percentage of patients with low disease activity at 24 weeks after randomization (CDAI) | At 36 weeks visit (corresponding to 24 weeks after randomization)
  Percentage of patients in low disease activity using definition : 2.8<CDAI≤10, at 24 weeks after randomization
Percentage of patients with low disease activity at 24 weeks after randomization (SDAI) | At 36 weeks visit (corresponding to 24 weeks after randomization)
  Percentage of patients in low disease activity using definition : 3.3<SDAI≤11, at 24 weeks after randomization
Percentage of patients with low disease activity at 36 weeks after randomization (DAS28-ESR) | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Percentage of patients in low disease activity using definition : 2.6≤DAS28-ESR≤3.2, at 36 weeks after randomization
Percentage of patients with low disease activity at 36 weeks after randomization (DAS28-CRP) | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Percentage of patients in low disease activity using definition : 2.6≤DAS28-CRP≤3.2, at 36 weeks after randomization
Percentage of patients with low disease activity at 36 weeks after randomization (CDAI) | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Percentage of patients in low disease activity using definition : 2.8<CDAI≤10, at 36 weeks after randomization
Percentage of patients with low disease activity at 36 weeks after randomization (SDAI) | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Percentage of patients in low disease activity using definition : 3.3<SDAI≤11, at 36 weeks after randomization
Proportion of responder patients at 12 weeks after randomization | At 24 weeks visit (corresponding to 12 weeks after randomization)
  Proportion of responders using EULAR (European Alliance of Associations for Rheumatology) definition (variations of DAS28-CRP from baseline >0.6 and DAS28-CRP≤5.1) at 12 weeks after randomization.
Proportion of responder patients at 24 weeks after randomization | At 36 weeks visit (corresponding to 24 weeks after randomization)
  Proportion of responders using EULAR definition (variations of DAS28-CRP from baseline >0.6 and DAS28-CRP≤5.1) at 24 weeks after randomization.
Proportion of responder patients at 36 weeks after randomization | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Proportion of responders using EULAR definition (variations of DAS28-CRP from baseline >0.6 and DAS28-CRP≤5.1) at 36 weeks after randomization.
Variations in the results of health assessment questionnaires administered to patients - HAQ-DI | Between baseline and 48 weeks
  Values and variations from baseline of patient-reported outcomes including health assessment questionnaire (HAQ-DI)
  The Health Assessment Questionnaire Disability Index (HAQ-DI) is an assessment of functional impairment. There are 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do).
Variations in the results of health assessment questionnaires administered to patients - EQ5D | Between baseline and 48 weeks
  Values and variations from baseline of patient-reported outcomes including health assessment questionnaire EQ5D
  The EuroQol 5-dimensional descriptive system (EQ5D) is a Health Assessment Scale quality of life questionnaire evaluating: mobility, washing and dressing, daily activities, pain and anxiety. Each question has 3 levels of answers: No problem, some problems and important problems.
Variations in the results of health assessment questionnaires administered to patients - SF-36 | Between baseline and 48 weeks
  Values and variations from baseline of patient-reported outcomes including health assessment questionnaire SF-36
  The Medical Outcomes Study 36-item Short-Form Health Survey (SF-36) is a patient-operated, self-administered measure created to assess health-related quality of life
Variation in autoantibody titers (RF) | between baseline and 48 weeks
  Variation of auto-antibodies titles (RF (rheumatoid factor)) and correlation of these variations with remission rate defined by DAS28-CRP<2.6.
Variation in autoantibody titers (ACPA) | between baseline and 48 weeks
  Variation of auto-antibodies titles (ACPA (Anti Citrullinated Peptides Antibodies)) and correlation of these variations with remission rate defined by DAS28-CRP<2.6.
Frequency of flares | between baseline and 48 weeks
  Frequency of flares assessed using the FLARE questionnaire completed by the patient between visits
  The self-administered Flare Assessment in Rheumatoid Arthritis (FLARE) is a self-administered questionnaire that was developed to help identify patients who had flare in the interval between 2 rheumatology consultations.
Cumulative doses of steroids consumed | between baseline and 48 weeks
  Cumulative doses of steroids collected with a booklet between baseline and 48 weeks
Percentage of Serious Adverse Events Occurring | between baseline and 48 weeks
  Safety: rates of serious adverse events including severe infections between baseline and 48 weeks
Variation of medical costs on Quality Adjusted Life Year | between baseline and 48 weeks
  Cost efficacy analysis based on direct and indirect costs and QALY (Quality Adjusted Life Year) between baseline and 48 weeks.
Variation of Sharp's score | between baseline and 48 weeks
  Variations Sharp's score between baseline and 48 weeks
  The Sharp method for scoring radiographs of hands and feet in rheumatoid arthritis.
  The method includes, in each hand, 16 areas for erosions and 15 areas for joint space narrowing, and, in each foot, 6 areas for erosions and 6 areas for joint space narrowing.
  The maximal erosion score for each hand is thus 80, considering the 16 areas for erosions per hand.
  Maximal total narrowing/(sub)luxation score in the hands is 120. Maximal total erosion score (hands and feet) is 280. Maximal total narrowing/(sub)luxation score in the feet is 48. Maximal total narrowing/(sub)luxation score (hands and feet) is 168.
  Maximal total Sharp score is 448.
  Sharp score will be calculated at W0 (baseline) and W48 (last visit). Variation of Shard score= score at W48- score at W0.
Percentage of patients remaining on abatacept | At 48 weeks visit (corresponding to 36 weeks after randomization)
  Percentage of patients remaining on abatacept in the sequential arm and on the 1st TNF inhibitor in the control arm at 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacques MOREL, MD-PhD, Study Director — UF of Montpellier
Locations (17):
- France (16):
  - Centre Hospitalier Universitaire de Montpellier, Montpellier, France
  - CHU Bordeaux groupe Pellegrin, Bordeaux
  - CHU de Brest La Cavale Blanche, Brest
  - Centre Hospitalier de Cahors, Cahors
  - CHD Vendée, La Roche-sur-Yon
  - CH du Mans, Le Mans
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU de Nîmes Carémeau, Nîmes
  - CHR Orléans Nouvel hôpital d'Orléans, Orléans
  - APHP Bicêtre, Paris
  - APHP Cochin, Paris
  - APHP La Pitié Salpetrière, Paris
  - CHU de Strasbourg Hautepierre, Strasbourg
  - Chu Purpan, Toulouse
  - CHU de Tours - Hopital Trousseau, Tours
- Centre hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: Undecided